CLINICAL TRIAL: NCT01487681
Title: Prevaccination Distribution of Cervical Human Papillomavirus (HPV) Types and Their Associations With Invasive Cervical Cancer and Its Precursors in Yangtze River Delta Area, China
Brief Title: Prevaccination Study of Cervical Human Papillomavirus Types in Yangtze River Delta Area, China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xing Xie, MD (Other)
Responsible Party: Sponsor-Investigator, Xing Xie, MD, Professor of Obstetrics and Gynecology，Director of Women's hospital, School of medicine, Zhejiang University, Zhejiang University
Organization: Zhejiang University (Other)
Other Study IDs: IISP 40192
Record Dates: First submitted 2011-11-30; First posted 2011-12-07 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-12

CONDITIONS: Human Papilloma Virus; Cervical Cancer; Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — The biospecimens are remainder tissue and exfoliated cervical cells of standard diagnosis and surgery.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Invasive cervical cancer
- Cervical intraepithelial neoplasia 2/3
- Cervical intraepithelial neoplasia 1

SUMMARY:
Human papilloma virus (HPV) infection contributes as a main causative factor to the development of invasive cervical cancer (ICC) and its precursors (cervical intraepithelial neoplasia, CIN). Currently, two prophylactic vaccines are employed for the prevention of genital HPV infection. As the prophylactic efficacy is type-restricted, determining the type-specific HPV distribution and their associations with ICC and its precursors would provide essential information in assessment of HPV vaccination program impact. The baseline information is also important for monitoring possible changes in type-specific HPV distribution after vaccination has been introduced.

Prevalence of HPV infection varies considerably across the world, and data were limited from less-developed countries. Knowledge of the detail pattern of HPV type-specific distribution in each region will be essential for public health policy decisions. This will also form the basis for determining which types should be included in future generation HPV vaccines targeted to specific regions.

While most studies were focus on ICC and high-grade cervical lesions, the association between HPV types and the progression of CIN1 has rarely been studied. CIN1 is an insensitive histopathological sign of HPV infection, most of which will spontaneously regress to normal with host immune system. However, some genotypes have been described as being more persistent and associated with progression from low-grade lesions to high-grade lesions, even ICC. Geographical data on type-specific prevalence of HPV in CIN1 with appropriately designed prospective studies would be helpful in identifying types preferentially associated with progression to malignancy and accurately predicting the future impact of vaccination in specific regions.

Free vaccination supported by the government appears to be unlikely at present in China. Thus, individuals need to pay the cost of vaccines for themselves presently. Yangtze River Delta Area is the most economically developed regions in China, and people here may become the largest vaccinated population at their own expense in China. To the best of the investigators knowledge, no multi-center study on HPV type-specific distribution and their associations with ICC and its precursors is available in Yangtze River Delta Area, China, which highlights the need for timely study in this region before large scale vaccination programs are carried out.

DETAILED DESCRIPTION:
The incidence of cervical cancer estimated to be 500,000 cases per year with a 50% case fatality rate. Human papilloma virus (HPV) infection, which is the most common sexually transmitted viral infection, contributes as a main causative factor to the development of invasive cervical cancer (ICC) and its precursors (cervical intraepithelial neoplasia, CIN). Thus, prophylactic HPV vaccines hold great promise to reduce the global burden of cervical cancer, especially in areas with no or limited screening.

Currently, two prophylactic vaccines, a quadrivalent (Gardasil®, Merck & Co. Inc) and a bivalent (Cervarix™, GlaxoSmithKline) vaccine, are employed for the prevention of genital HPV infection in more than 100 countries, and showed high efficacy for the prevention of target HPV related CIN2+. Merck is also conducting a Phase III trial of a vaccine protecting against nine types. As the prophylactic efficacy is type-restricted and not all the different types of HPV are covered by currently available vaccines, determining the type-specific HPV distribution and their associations with ICC and its precursors would provide essential information in assessment of HPV vaccination program impact. What is more, it is possible that the decrease in the prevalence of the target types of these vaccines could affect the distribution of other types, so the baseline information is also important for monitoring possible changes in type-specific HPV distribution after vaccination has been introduced.

Previous meta-analyses had showed that in ICC, HPV 16 was most common, followed by HPV 18, while HPV 16/18 prevalence was 52% among high-grade cervical lesions. However, the prevalence of HPV infection varies considerably across the world, and data were limited from less-developed countries, let alone multi-center studies. Knowledge of the detail pattern of HPV type-specific distribution in each region will be essential for public health policy decisions. This will also form the basis for determining which types should be included in future generation HPV vaccines targeted to specific regions. A tailed HPV vaccine according to regional prevalence would best serve the population in primary prevention for ICC.

On the other side, while most studies were focus on ICC and high-grade cervical lesions, the association between HPV types and the progression of CIN1 has rarely been studied. CIN1 is an insensitive histopathological sign of HPV infection, most of which will spontaneously regress to normal with host immune system. However, some genotypes have been described as being more persistent and associated with progression from low-grade lesions to high-grade lesions, even ICC. Geographical data on type-specific prevalence of HPV in CIN1 with appropriately designed prospective studies would be helpful in identifying types preferentially associated with progression to malignancy and accurately predicting the future impact of vaccination in specific regions.

Recently, a randomized, double-blind trial testing the safety and efficacy of the quadrivalent vaccine (Gardasil®, Merck & Co. Inc) in Chinese women (V501-041-00) has been conducting and is proposed to be finished in three years. The bivalent vaccine (Cervarix™, GlaxoSmithKline) also has applied the phase III double-blind, randomized controlled trial in Chinese women. These prophylactic vaccines might be licensed and commercially available in China after trials finish. However, free vaccination supported by the government appears to be unlikely at present according to current economic status of China. Thus, individuals at least presently need to pay the cost of vaccines for themselves.

Yangtze River Delta Area, including Shanghai city, Zhejiang Province and Jiangsu Province, is the most economically developed regions in China. According to media report, the total GDP in Yangtze River Delta area was approximated 1.064 trillion U.S. dollars in 2010, and the per capita GDP has exceeded 4,000 U.S. dollars since 2005. As people here have the highest health awareness and needs, they may become the largest vaccinated population at their own expense in China. To the best of our knowledge, no multi-center study on HPV type-specific distribution and their associations with ICC and its precursors is available in Yangtze River Delta Area, China, except for the mono-center study in Zhejiang Province, which highlights the need for timely study in this region before large scale vaccination programs are carried out.

ELIGIBILITY:
Inclusion Criteria:

* Women with histologically confirmed CIN1, CIN2, CIN3 or invasive cervical cancer (ICC)

Exclusion Criteria:

* Women with a history of immunodeficiency disorders, including HIV, and those who had undergone chemoradiotherapy for cervical cancer were excluded.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with histologically confirmed CIN1, CIN2, CIN3 or invasive cervical cancer (ICC)
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of each HPV type in patients with invasive cervical cancer, cervical intraepithelial neoplasia 2-3 and cervical intraepithelial neoplasia 1, respectively, in Yangtze River Delta Area, China | One year

SECONDARY OUTCOMES:
HPV types significantly associated with persistence or progression of cervical intraepithelial neoplasia 1 at one year in Yangtze River Delta Area, China | One year

CONTACTS AND LOCATIONS:
Overall Officials: Xing Xie, Professor, Study Director — Women's Hospital School Of Medicine Zhejiang University
Locations (1):
- Women's hospital, School of medicine, Zhejiang University, Hangzhou, Zhejiang, China